CLINICAL TRIAL: NCT06837363
Title: A Multicenter Confirmation Clinical Trial of Untact Upper Extremity Rehabilitation Using Smart Board for Late Subacute and Chronic Patients With Brain Disorder - a Randomized Single-blinded Controlled Trial
Brief Title: Effect of Untact Upper Extremity Rehabilitation Using a Smart Board for Late Subacute and Chronic Patients With Brain Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-09-105
Record Dates: First submitted 2025-01-13; First posted 2025-02-20 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Home Based Rehabilitation; Brain Disorder
MeSH Terms: conditions — Brain Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Neofect Smart Board (Experimental): home-based upper limb rehabilitation training using the Neofect Smart board
  Interventions: Device: Home-based Neofect Smart board
- home-based occupational therapy (Active Comparator): home-based upper limb rehabilitation training using the workbook provided by the research team
  Interventions: Other: home-based occupational therapy

INTERVENTIONS:
Device: Home-based Neofect Smart board — a total of 20 sessions of home-based upper limb rehabilitation training using the Neofect Smart board, with 30 minutes per session, 1 session per day, 5 days a week, for 4 weeeks.
  Arms: Home-based Neofect Smart Board
Other: home-based occupational therapy — a total of 20 sessions of home-based upper limb rehabilitation training using the workbook provided by the research team , with 30 minutes per session, 1 session per day, 5 days a week, for 4 weeeks.
  Arms: home-based occupational therapy

SUMMARY:
The aim is to clinically validate the clinical efficacy, usability, and safety of home-based upper limb rehabilitation training using the Neofect Smart Board by comparing the effects between a group using the home-based Neofect Smart Board and a group performing conventional home-based occupational therapy in patients with upper limb dysfunction in the late subacute and chronic stages of neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neurological diseases aged 19 to 85 years old
* Patients with hemiparesis lasting for more than 3 months due to neurological diseases (stroke, traumatic brain injury, brain tumor) and impaired upper limb function
* Patients with shoulder flexor and adductor muscle strength of MRC grade 2 or higher
* Patients with shoulder extensor and abductor spasticity of MAS grade 1+ or lower
* Participants with sufficient cognitive function to understand the instructions from the researcher and the smart board, and to perform the tasks (K-MMSE ≥21)

Exclusion Criteria:

* pre-existing significant neurogenic disorders
* major psychiatric disorders such as schizophrenia, bipolar disorder, or dementia
* History of diseases that caused pain or muscle atrophy in the affected upper limb before the onset of the neurological disease, which interfered with rehabilitation
* Severe spasticity of the affected upper limb (Modified Ashworth Scale score ≥3)
* skin disorders or open wounds on the affected upper limb
* Amputation, fractures, or soft tissue-related diseases or injuries on the affected upper limb
* severe pain that interferes with rehabilitation of the affected upper limb (Numeric Rating Scale > 6)
* Inability to maintain a seated posture for more than 10 minutes, which is required for using the smart board
* Significant visual impairment to the extent that the screen cannot be recognized when using the smart board

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of uper limb score in Fugl-Meyer assessment | Within 14 days before the intervention, within 2 days after intervention
  (upper limb motor score in Fugl-Meyer assessment at post-intervention) - (upper limb motor score in Fugl-Meyer assessment at baseline) Higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung medical center, Seoul, South Korea